CLINICAL TRIAL: NCT00887900
Title: Deep Anterior Lamellar Keratoplasty by Big-Bubble Technique: Results and Complications
Brief Title: Deep Anterior Lamellar Keratoplasty (DALK)
Acronym: DALK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Responsible Party: PATRICK TZELIKIS, HOB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DALK
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Keratoconus
Keywords: lamellar keratoplasty; keratoconus; penetrated keratoplasty; Visual acuity
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Submitted to deep anterior lamellar keratoplasty (DALK) using the big-bubble technique.
  Interventions: Procedure: Deep anterior lamellar keratoplasty (DALK)
- 2 (Active Comparator): Submitted to regular penetrating keratoplasty
  Interventions: Procedure: Penetrated keratoplasty

INTERVENTIONS:
Procedure: Deep anterior lamellar keratoplasty (DALK) — Deep anterior lamellar keratoplasty (DALK) using the big-bubble technique.
  Other Names: GROUP 1: DALK
  Arms: 1
Procedure: Penetrated keratoplasty — Regular corneal transplant using the penetrated keratoplasty technique
  Other Names: GROUP 2: PK
  Arms: 2

SUMMARY:
The purpose of this study is to report outcomes of deep anterior lamellar keratoplasty (DALK) using the big-bubble technique.

DETAILED DESCRIPTION:
Purpose: To report outcomes of deep anterior lamellar keratoplasty (DALK) using the big-bubble technique.

Methods: Thirty four unselected consecutive patients were submitted to DALK big-bubble technique. Intraoperative and postoperative complications, postoperative uncorrected visual acuity (UCVA), best spectacle-corrected visual acuity (BSCVA), spherical equivalent (SE), corneal topography, and endothelial cell density were evaluated. All patients were followed for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* keratoconus

Exclusion Criteria:

* central endothelial cell count less than 2000 cells/mm2
* glaucoma or intraocular pressure greater than 21 mmHg
* amblyopia
* retinal abnormalities
* diabetes mellitus
* steroid or immunosuppressive treatment
* connective tissue diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To report outcomes of deep anterior lamellar keratoplasty (DALK) using the big-bubble technique. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: PATRICK F TZELIKIS, PhD, MD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital Oftalmologico de Brasília, Brasília, Federal District, Brazil

REFERENCES:
- [Result] Tan DT, Parthasarathy A. Deep anterior lamellar keratoplasty for keratoconus. Cornea. 2007 Sep;26(8):1025; author reply 1025-6. doi: 10.1097/ICO.0b013e31805771e3. No abstract available. PMID 17721317
- [Result] Vajpayee RB, Tyagi J, Sharma N, Kumar N, Jhanji V, Titiyal JS. Deep anterior lamellar keratoplasty by big-bubble technique for treatment corneal stromal opacities. Am J Ophthalmol. 2007 Jun;143(6):954-957. doi: 10.1016/j.ajo.2007.02.036. Epub 2007 Apr 16. PMID 17434435
- [Result] Ardjomand N, Hau S, McAlister JC, Bunce C, Galaretta D, Tuft SJ, Larkin DF. Quality of vision and graft thickness in deep anterior lamellar and penetrating corneal allografts. Am J Ophthalmol. 2007 Feb;143(2):228-235. doi: 10.1016/j.ajo.2006.10.043. Epub 2006 Nov 30. PMID 17258522
- [Derived] Tzelikis PF, Santos JD, Garcez RC, Akaishi L. [Deep anterior lamellar keratoplasty by big-bubble technique]. Arq Bras Oftalmol. 2011 Nov-Dec;74(6):435-40. doi: 10.1590/s0004-27492011000600011. Portuguese. PMID 22331118
- See also: PUBMED — http://www.ncbi.nlm.nih.gov/pubmed